CLINICAL TRIAL: NCT05586581
Title: PET Imaging of Synaptic Density Combined With Neuroimmunologic Measures to Reveal Mechanisms of HIV Neuropathogenesis During ART
Brief Title: SV2A & TSPO PET Imaging Measures to Reveal Mechanisms of HIV Neuropathogenesis During Antiretroviral Therapy
Acronym: ART
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Serena Spudich, MD, Gilbert H. Glaser Professor of Neurology, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000033582; 5R01MH125396 (NIH)
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: HIV Associated Neurocognitive Disorder; HIV Dementia; HIV Encephalitis; Healthy
Keywords: Human immunodeficiency virus; Positron-Emission Tomography Imaging; Magnetic Resonance Imaging; Cerebrospinal Fluid; SV2A PET; TSPO PET; Neuro-immune dysfunction; Neuro-Inflammation; Biomarkers of inflammation; Neuronal Injury; Neurocognitive functioning; Hippocampus; Microglia; Neuropathogenesis; antiretroviral therapy
MeSH Terms: conditions — AIDS Dementia Complex; Acquired Immunodeficiency Syndrome | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one; (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Intervention Model Description: In this study, people living with treated suppressed HIV infection (PLWH) and matched HIV-negative controls will be scanned using anatomical magnetic resonance imaging (MRI) and PET. All participants will receive two SV2A PET scans (baseline and 2 years). A subset of PLWH participants will be asked to complete a TSPO PET scan on the same day as the baseline SV2A PET scan. Participants will undergo phlebotomy and medical/mental health and substance use histories for eligibility, and may also complete an ECG, blood tests, an optional lumbar puncture, neurocognitive testing & behavioral/mood questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- People living with treated suppressed HIV infection (PLWH) (Experimental): 40 PLWH participants will be scanned using anatomical magnetic resonance imaging (MRI) and undergo two SV2A (11C-UCB-J) PET scans with arterial sampling and full radio metabolite analysis to obtain measures of synaptic density at baseline and 24 months (2 years). For each SV2A PET, up to 20 millicurie (mCi) of [11C], UCB-J will be administered by an intravenous line (IV) with a scan duration of up to 120 minutes.
  A subset of PLWH (n=20) will participate in TSPO (11C-PBR28) PET scans on the same day as the baseline SV2A PET scan. For a TSPO PET, up to 20 mCi of [11C], PBR28 will be administered by an intravenous line (IV) with a scan duration of up to 120 minutes.
  Interventions: Drug: SV2A PET; Drug: TSPO PET
- HIV-Negative Control (HIV-) (Experimental): 30 HIV-Negative Control (HIV-) participants will be scanned using anatomical magnetic resonance imaging (MRI) and undergo two SV2A (11C-UCB-J) PET scans with arterial sampling and full radio metabolite analysis to obtain measures of synaptic density at baseline and 24 months (2 years). For each SV2A PET, up to 20 mCi of [11C], UCB-J will be administered by an intravenous line (IV) with a scan duration of up to 120 minutes.
  Interventions: Drug: SV2A PET

INTERVENTIONS:
Drug: SV2A PET — SV2A PET scan with radiotracer [11C]UCB-J for imaging synaptic density in the brain
  Other Names: [11C]UCB-J; [11C]APP311
Drug: TSPO PET — TSPO PET scan with radiotracer [11C]PBR28 for imaging of neuroimmune status
  Other Names: [11C]PBR28
  Arms: People living with treated suppressed HIV infection (PLWH)

SUMMARY:
The purpose of this study is to longitudinally characterize and evaluate changes in synaptic density in the brain using novel positron-emission tomography (PET) scans; magnetic resonance imaging (MRI), and clinical laboratory markers associated with HIV-related injury in the central nervous system. This study will test hypotheses relating to the presence and mechanisms of aberrant brain structure at the synaptic level in living humans with virologically controlled HIV on antiretroviral therapy. To evaluate associations between PET imaging radiotracers [11C]UCB-J, a ligand for presynaptic vesicle protein 2A (SV2A), a vesicle membrane protein expressed in synapses, and PET [11C]PBR28 a measure of microglia function in the brain, the Yale PET center has developed an advanced approach of combining multiple distinct ligands in coordinated same-day PET imaging. Additionally, the study will evaluate the associations of this novel synaptic density marker with well-established clinical measures of neurocognitive performance and laboratory measures of blood and cerebrospinal fluid (CSF).

DETAILED DESCRIPTION:
The HIV PET plus study builds upon the compelling preliminary findings of the investigators HIV PET pilot study (Yale Internal Review Board (IRB) #2000024620) that brain SV2A PET successfully identifies regions of reduced synaptic density, including a hippocampal-frontostriatal neural circuit that is relevant to central nervous system (CNS) dysfunction in PLWH on ART

The primary aims of this study are as follows:

Aim 1. To evaluate cross-sectional differences and 24-month longitudinal changes in synaptic density in PLWH on suppressive ART relative to matched HIV-negative (HIV-) controls. Synaptic density will be measured with SV2A PET scans acquired at baseline and two years in 40 PLWH on ART and in 30 HIV-, matched for age, gender, ethnicity, and history of substance use.

Hypotheses: (1a) Synaptic density in a hippocampal-frontostriatal neural circuit will be reduced in PLWH relative to matched HIV-; (1b) Synaptic density in this circuit will decline at a greater rate in PLWH relative to HIV-.

Aim 2. To determine, in PLWH on ART, the extent to which microglia levels impact synaptic density. Microglia levels will be measured with TSPO PET scans concurrently acquired with SV2A PET scans in a subset of 20 PLWH from Aim 1 at baseline, followed by repeat SV2A PET scans at 24 months.

Hypotheses: (2a) Greater microglia levels in a hippocampal-frontostriatal circuit will be associated with decreased synaptic density in this circuit; and (2b) Greater microglial levels at baseline will be a longitudinal predictor of a greater decline in synaptic density in this neural circuit over 24 months.

Aim 3. To determine the role of synaptic density in mediating the relation between microglia level, laboratory biomarkers of inflammation and neuronal injury, and neurocognitive functioning in PLWH. Blood, cerebrospinal fluid, and neurocognitive measures will be acquired in 40 PLWH on ART at baseline and 2 years with SV2A PET. The investigators will use parallel processing statistical approaches to examine multimodal longitudinal associations between baseline microglial activation, and changes in synaptic density, laboratory biomarkers and neurocognitive functioning to understand the molecular neuropathogenesis of CNS impairment in PLWH on ART.

Hypothesis: (3) In PWLH on ART, greater hippocampal-frontostriatal microglial activation at baseline will be associated with greater 24-month reductions in synaptic density, which will in turn be associated with greater reductions in neurocognitive functioning, particularly on measures of learning and memory.

ELIGIBILITY:
PLWH Inclusion Criteria:

* Voluntary, written, informed consent (signed and dated)
* For females, a negative urine or serum pregnancy (HCG) test at screening and on each scan day before initiation of any scan procedures.
* HIV infection on cART with documented viral suppression for at least one year. Plasma viral suppression will be defined as no more than one viral load
* Test above 20 HIV RNA cps/mL in the year prior to screening and no HIV RNA tests above 200 cps/mL in the same span.
* Willingness to participate in MRI, PET, phlebotomy, and Neuropsychological Testing (NPT) Assessments & Surveys.

PLWH Exclusion Criteria:

* Active substance dependence (e.g., heroin, alcohol, cocaine, sedative hypnotics, methamphetamine) as determined by the standardized Behavioral Assessments.
* A history of significant non-HIV related neurological illness (e.g., cerebrovascular, seizures, traumatic brain injury).
* Medical contraindications to the administration of radioactivity (e.g., prior radiation exposure within the past year from research, or from workplace exposure, that in combination with the planned scans would exceed the FDA limit for annual radiation exposure).
* Medical contraindications to participation in a magnetic resonance imaging procedure (e.g., ferromagnetic implants/foreign bodies, claustrophobia, cardiac pacemaker, prosthetic valve, otologic implant, etc.).
* History of a bleeding disorder, low platelet count, or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto).

HIV - Inclusion Criteria:

* Voluntary, written, informed consent (signed and dated)
* For females, a negative urine or serum pregnancy (HCG) test at screening and on each scan day before initiation of any scan procedures.
* Willingness to participate in phlebotomy, NPT Assessments & Surveys, MRI, and PET.
* Physically healthy by medical history, physical, neurological, and laboratory examinations, as judged by the principal investigator.
* Have a negative test for HIV on file within the last three months or willing to have an HIV test in the current study.

HIV- Exclusion Criteria:

* Active substance dependence (e.g., heroin, alcohol, cocaine, sedative hypnotics, methamphetamine) as determined by the standardized Behavioral Assessments.
* A history of significant neurological illness (e.g., cerebrovascular, seizures, traumatic brain injury).
* Medical contraindications to the administration of radioactivity (e.g., prior radiation exposure within the past year, from research, or from workplace exposure, that in combination with the planned scans would exceed the FDA limit for annual radiation exposure)
* Medical contraindications to participation in a magnetic resonance imaging procedure (e.g., ferromagnetic implants/foreign bodies, claustrophobia, cardiac pacemaker, prosthetic valve, otologic implant, etc.
* History of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure for 11C-UCB-J will be the binding potential of 11C-UCB-J, specifically non-displaceable binding potential (BPND), the ratio of the specifically bound radioligand to that of nondisplaceable radioligand in tissue. | Through study completion date, an average of 5 years.
  Preliminary data from the investigators' pilot study revealed SV2A PET imaging with radiotracer 11C-UCB-J identified regions of reduced synaptic density in suppressed PLWH compared to matched HIV-negative controls.
  PET and MRI imaging data will be processed for quantification of 11C-UCB-J imaging data in a larger group of suppressed PLWH compared to matched HIV-negative controls to test-retest reproducibility of 11C-UCB-J.
Change in cross-sectional differences and 24-month longitudinal changes in synaptic density in PLWH on suppressive ART relative to matched HIV-negative controls | Baseline and 24 months
  Baseline and 24 Month PET and MRI imaging data will be processed for a linear mixed-effects model (LMM) to compare changes in hippocampal-frontostriatal 11C-UCB-J BPND between PLWH and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Spudich, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicne, Neuro ID Research Program, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No